CLINICAL TRIAL: NCT05695989
Title: Prospective, Multi-center, Single-arm, Open Label Study Designed to Assess the Safety and Feasibility of the Use of the Dual Robotic Arm Accessory With the Levita Magnetic Surgical System in Laparoscopic Procedures
Brief Title: Safety and Feasibility of the Use of the Dual Robotic Arm Accessory With the Levita Magnetic Surgical System in Laparoscopic Procedures
Acronym: MARS GI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Levita Magnetics (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP008
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Bariatric Surgery Candidate; Cholelithiases; Other Disease
MeSH Terms: conditions — Cholelithiasis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DRAA (Dual Robotic Arm Accessory) (Experimental): Levita has developed a Robotic Platform (DRAA) to assist in external management of the controlling magnet and the laparoscopic camera, which would give better control of surgical tools to the surgeon.
  Interventions: Device: Dual Robotic Arm Accessory (DRAA)

INTERVENTIONS:
Device: Dual Robotic Arm Accessory (DRAA) — Dual Robotic Arm Accessory (DRAA)

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of the Levita Dual Robotic Arm Accessory (DRAA) used with the Levita Magnetic Surgical System (MSS)

DETAILED DESCRIPTION:
Prospective, multi-center, single-arm, open label study designed to assess the safety and feasibility of the use of the Dual Robotic Arm Accessory with the Levita Magnetic Surgical System in laparoscopic procedures

ELIGIBILITY:
Inclusion Criteria:

* • Subject is at least 18 years of age

  * Subject is scheduled to undergo elective laparoscopic procedure
  * Subject signs a written Informed Consent Form (ICF) to participate in the study prior to any study required procedures

Exclusion Criteria:

* • Subjects with pacemakers, defibrillators, or other electromedical implants

  * Subjects with ferromagnetic implants
  * Subjects with significant comorbidities: cardiovascular, neuromuscular, chronic obstructive pulmonary disease, and urological disease (renal failure)
  * Subjects with a clinical history of impaired coagulation confirmed by abnormal blood tests
  * Subject has an anatomical abnormality or disease of intended target tissue noted after initiation of index procedure that would prevent device use
  * Subject is pregnant or wishes to become pregnant during the length of study participation
  * Subject is not likely to comply with the follow-up evaluation schedule
  * Subject is participating in a clinical trial of another investigational drug or device Prisoner or under incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Jimenez, MD, Principal Investigator — Hospital Tisne
Locations (3):
- Chile (3):
  - Hospital Tisne, Santiago, Santiago Metropolitan
  - Clinica Colonial, Santiago
  - Hospital Fach, Santiago

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DRAA (Dual Robotic Arm Accessory)
Started | 22
Completed | 20
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | DRAA (Dual Robotic Arm Accessory)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Chile | 20

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events- Safety
Description: Adverse events related to the device
Time Frame: 30 days
Measure: Number; unit: Device related adverse events
Arm/Group | DRAA (Dual Robotic Arm Accessory)
Number analyzed (Participants) | 20
Device related adverse events | 0

2. Secondary Outcome: Rate That the Dual Robotic Arm Accessory (DRAA) is Able to Engage, Move, and Decouple With the Magnetic Surgical System as Controlled by the Surgeon
Description: Ratio of successful attempts vs unsuccessful attempts
Time Frame: Surgery time
Measure: Number; unit: Number Surgeries completed successfully
Arm/Group | DRAA (Dual Robotic Arm Accessory)
Number analyzed (Participants) | 20
Number Surgeries completed successfully | 20

3. Secondary Outcome: Conversion Rate to Open Surgery
Description: Ratio of conversion from laparoscopic to open surgery due to inability of the robotic system to provide adequate visualization
Time Frame: Surgery time
Measure: Number; unit: Converted procedures
Arm/Group | DRAA (Dual Robotic Arm Accessory)
Number analyzed (Participants) | 20
Converted procedures | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE) and serious adverse events (SAEs) were recorded from index procedure through study exit (30 day follow up).
Arm/Group | DRAA (Dual Robotic Arm Accessory)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 12/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DRAA (Dual Robotic Arm Accessory) (N=20)
Allergic Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis in surgical wound (Skin and subcutaneous tissue disorders) | 3 (3)
Liver capsule minor abrasion without clinically relevant concern (Surgical and medical procedures) | 3 (3)
Petechia (Skin and subcutaneous tissue disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT05695989/Prot_SAP_000.pdf